CLINICAL TRIAL: NCT06770582
Title: Randomized Phase II Trial of Pembrolizumab and Radiation vs. Radiation and Concurrent Chemotherapy for High-Grade T1 Bladder Cancer (PARRC Trial)
Brief Title: Testing the Addition of the Immunotherapy Drug, Pembrolizumab, to Radiation Therapy Compared to the Usual Chemotherapy Treatment During Radiation Therapy for Bladder Cancer, PARRC Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-00008; NCI-2025-00008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU014 (Other: NRG Oncology); NRG-GU014 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Non-Muscle Invasive Bladder Urothelial Carcinoma; Recurrent Non-Muscle Invasive Bladder Urothelial Carcinoma; Stage I Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Gemcitabine; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex; pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Chemotherapy and radiation) (Active Comparator): Patients receive one of the following chemotherapy regimens per physicians choice: 1) cisplatin IV once per week for 4 weeks, 2) gemcitabine IV on days 1, 4, 8, 11, 15, 18, 22, and 25, or 3) mitomycin IV on day 1 and 5-fluorouracil IV continuously over 120 hours on days 1-5 and 16-20. Patients receiving cisplatin or gemcitabine continue chemotherapy for 6 weeks if they are receiving radiation according to the standard hypofractionated radiation schedule. Starting on day 1, patients also receive radiation therapy for 20, 32, or 36 treatments over 4-7 weeks. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo CT/MRI and blood sample collection throughout the study. Patients may also undergo optional urine sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm 2 (Pembrolizumab and radiation) (Experimental): Patients receive pembrolizumab IV over 25-40 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for 9 cycles in the absence of disease progression or unacceptable toxicity. Starting on day 1, patients also receive radiation therapy for 20, 32, or 36 treatments over 4-7 weeks. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo CT/MRI and blood sample collection throughout the study. Patients may also undergo optional urine sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm 1 (Chemotherapy and radiation)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm 1 (Chemotherapy and radiation)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm 1 (Chemotherapy and radiation)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Given IV
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
  Arms: Arm 1 (Chemotherapy and radiation)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm 2 (Pembrolizumab and radiation)
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II trial compares the use of pembrolizumab and radiation therapy to chemotherapy with cisplatin, gemcitabine, 5-fluorouracil or mitomycin-C and radiation therapy for the treatment of non-muscle invasive bladder cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as cisplatin, gemcitabine, 5-fluorouracil or mitomycin-C, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Giving pembrolizumab with radiation may kill more tumor cells than chemotherapy with radiation therapy in patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare bladder-intact event-free survival.

SECONDARY OBJECTIVES:

I. To assess complete response by cystoscopy at 6 months. II. To assess disease-free survival. III. To assess local-regional control. IV. To assess metastasis-free survival. V. To assess overall survival. VI. To assess quality of life using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and the Bladder Cancer Index at 18 months.

VII. To assess Common Terminology Criteria for Adverse Events (CTCAE) adverse events (both acute and late).

EXPLORATORY OBJECTIVES:

I. To assess fatigue using the Patient Reported Outcomes Measurement Information System Fatigue-4A (PROMIS-Fatigue-4a).

II. To assess quality adjusted survival using European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L).

III. To assess cumulative quality of life using EORTC QLC-C30 and Bladder Cancer Index at 24 months.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive one of the following chemotherapy regimens per physicians choice: 1) cisplatin intravenously (IV) once per week for 4 weeks, 2) gemcitabine IV on days 1, 4, 8, 11, 15, 18, 22, and 25, or 3) mitomycin IV on day 1 and 5-fluorouracil IV continuously over 120 hours on days 1-5 and 16-20. Patients receiving cisplatin or gemcitabine continue chemotherapy for 6 weeks if they are receiving radiation according to the standard hypofractionated radiation schedule. Starting on day 1, patients also receive radiation therapy for 20, 32, or 36 treatments over 4-7 weeks. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT)/magnetic resonance imaging (MRI) and blood sample collection throughout the study. Patients may also undergo optional urine sample collection on study.

ARM 2: Patients receive pembrolizumab IV over 25-40 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for 9 cycles in the absence of disease progression or unacceptable toxicity. Starting on day 1, patients also receive radiation therapy for 20, 32, or 36 treatments over 4-7 weeks. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo CT/MRI and blood sample collection throughout the study. Patients may also undergo optional urine sample collection on study.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of T1 high-grade non-muscle invasive urothelial carcinoma of the bladder without radiographic evidence of regional nodal disease or metastatic disease (N0, M0) on CT, MRI, or positron emission tomography (PET)/CT scan who would otherwise be treated with cystectomy off-trial. Patients should have cystectomy recommended disease but do not need to be medically operable for a cystectomy to be eligible for the trial.

  * NOTE: Patients with nodal disease ≥ 1 cm on short-axis or with suspicious nodes that are PET-avid of any size are not eligible
* High grade T1 disease history that must meet at least ONE of the three criteria below:

  * Histologically confirmed recurrence with high-grade T1 urothelial carcinoma (+/- focal carcinoma in situ [CIS]) in the bladder following initial transurethral resection of bladder tumor (TURBT) and at least one induction course of intravesical therapy. Adequate induction course is defined as ≥ 5 doses of intravesical Bacillus Calmette-Guerin (BCG) or intravesical chemotherapy when BCG is not available.
  * T1 with pathologic high-risk features (lymphovascular invasion [LVI] or variant histology of micropapillary, sarcomatoid, or plasmacytoid features) post initial TURBT. (No prior intravesical therapy required)
  * Persistent high-grade T1 urothelial carcinoma at repeat TURBT (+/- focal CIS) in the bladder. (No prior intravesical therapy required)
* Restaging TURBT must be performed and must meet ALL of the following criteria below:

  * If there is absence of muscularis propria in the initial TURBT, there must be uninvolved muscularis propria in the restaging TURBT.
  * All grossly visible papillary tumors must be removed

    * Note: If the restaging TURBT is performed outside of the enrolling institution, an office cystoscopy should be performed by a Urologist who will be following the patient as part of the clinical trial
* No pure squamous cell carcinoma or adenocarcinoma of the bladder
* No neuroendocrine (small or large cell) features
* No diffuse carcinoma in situ determined on cystoscopy and biopsy (i.e. extensive carcinoma in situ that is not just tumor-associated CIS in the opinion of the site investigator)
* No prostatic urethral involvement
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy), tubal ligation or who is not postmenopausal
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 9 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 9 g/dl is acceptable)
* Adequate renal function defined as creatinine clearance (CrCL) of ≥ 30 mL/min by the Cockcroft-Gault formula, ≤ 1.5 × upper limit of normal (ULN) or creatinine levels > 1.5 × institutional ULN
* Total bilirubin ≤ institutional upper limit of normal (ULN) (Not applicable to patients with known Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* All adverse events of their most recent therapy/intervention must have resolved to < grade 3 or returned to baseline prior to registration
* No history of pelvic radiation therapy
* No prior systemic chemotherapy or immunotherapy for urothelial carcinoma. Prior treatment with local intravesical therapy including BCG or chemotherapy is allowed
* No prior treatment with anti-PD-1, anti PD-L1, anti PD-L2 or anti-CTLA4 antibody or any other antibody or drug targeting T-cell co-stimulation
* No live vaccine administered within 30 days of registration. All non live vaccines (including the coronavirus disease [COVID] vaccine) are allowed at any time during the study. Timing should minimize confusion with drug-related toxicities where possible
* Patients must have recovered from acute cardiac illness
* New York Heart Association Functional Classification II or better (New York Heart Association [NYHA] Functional Classification III/IV are not eligible) (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
* No active infection requiring IV antibiotics
* No active autoimmune disease that required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* No history of idiopathic pulmonary fibrosis, organizing pneumonia, (non-infectious) pneumonitis that required steroids or current pneumonitis
* No history of allogeneic bone marrow transplant or prior solid organ transplant
* No active tuberculosis
* No evidence of hydronephrosis
* No history of upper tract urothelial carcinoma within 24 months of registration
* No patients with a prior diagnosis of prostate cancer who have not received definitive treatment for their prostate cancer (e.g. on active surveillance)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* No glucocorticoids except physiologic doses are allowed. The use of doses of corticosteroids (defined as 10 mg prednisone or equivalent) is acceptable
* No history of allergic reaction to the drug excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2032-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Bladder intact event-free survival (BIEFS) | Up to 5 years
  Defined as time free of histologically proven recurrent T1-T4 recurrence, clinical evidence of nodal or distant metastasis, radical cystectomy (either for disease progression or due to toxicity), or death from any cause. Analysis will consist of estimation of the BIEFS curves via the Kaplan-Meier estimator and testing of the primary hypothesis using the stratified logrank test (one-sided). Additionally, the Cox proportional hazards model will be used to estimate the hazard ratio adjusting for stratification variables and any other baseline covariates that demonstrate any degree of imbalance by treatment arm.
Global quality of life | Up to 5 years
  Assessed using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC-QLQ-C30) global quality of life domain.

SECONDARY OUTCOMES:
Complete response by cystoscopy | At 6 months
  The proportion achieving complete response will be compared using the two-sample binomial test. Further analysis may consist of using a binary outcome regression model (i.e., logistic regression) to compute the relative odds of response adjusted for any factors that may appear imbalanced by treatment arm.
Disease free survival | Up to 5 years
  Defined in standard specification as time free of any disease failure (local/regional/distant), or death from any cause. Will be evaluated via the Kaplan-Meier estimator and logrank test.
Local-regional control | Up to 5 years
  Will be estimated via the cumulative incidence estimator, treating death as a competing event.
Metastasis free survival | Up to 5 years
  Will be evaluated via the Kaplan-Meier estimator and logrank test.
Overall survival | Up to 5 years
  Will be estimated via the Kaplan-Meier estimator.
Quality of life | Up to 2 years
  Assessed using the Bladder Cancer Index and EORTC-QLQ-C30.
Incidence of adverse events (AE) | Up to 3 years
  Assessed using the Common Terminology Criteria for Adverse Events. Counts and frequencies will be reported for the worst grade per AE experienced per patient by treatment arm. Differences in frequency by treatment arm of AE grade, singly or grouped into larger categories (for example, grade 3 or higher vs lower) with be tested using a chi-squared test or Fisher's exact test with a significance level of 0.05.
Bladder specific quality of life | Up to 2 years
  Using the Bladder Cancer Index.

OTHER OUTCOMES:
Quality adjusted survival | Up to 2 years
  Index scores from the European Quality of Life Five Dimension Five Level Scale will be calculated at each time point and change from baseline to post-treatment scores compared between treatment arms using a t-test with a 2-sided significance level of 0.05. If there are significant differences, then a quality-adjusted life year (QALY) analysis will be conducted. QALYs are defined by the weighted sum of different time episodes added up to a total quality-adjusted survival time. The difference in QALYs between arms will be reported along with the 95% confidence interval.
Fatigue | Up to 2 years
  Using Patient Reported Outcomes Measurement Information System Fatigue-4A. Calculated by summing all 4 questions (all 4 questions are required to be completed to score the tool). Raw scores range from 4 to 20 and are standardized to a T score following the scoring instructions.
Cumulative global quality of life | Up to 2 years
  Using the EORTC-QLQ-C30 and Bladder Cancer Index.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Baumann, Principal Investigator — NRG Oncology
Locations (107):
- United States (107):
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Shaw Cancer Center, Edwards, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Gonzales, Gonzales, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm